CLINICAL TRIAL: NCT01328951
Title: A Randomized, Double-Blind, Placebo-Controlled Phase III Study of First-Line Maintenance Tarceva Versus Tarceva at the Time of Disease Progression in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) Who Have Not Progressed Following 4 Cycles of Platinum-Based Chemotherapy
Brief Title: A Study of First-line Maintenance Erlotinib Versus Erlotinib at Disease Progression in Participants With Advanced Non-Small Cell Lung Cancer (NSCLC) Who Have Not Progressed Following Platinum-Based Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO25460
Record Dates: First submitted 2011-04-04; First posted 2011-04-05 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-06

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Early Erlotinib (Experimental): Participants will receive blinded erlotinib as 150 mg PO once daily in the maintenance setting until disease progression, death, or unacceptable toxicity. Those who demonstrate disease progression may be unblinded to receive an approved second-line therapy (but not EGFR targeted therapies) until disease progression, death, or unacceptable toxicity. Participants may be observed during a final SFU period after discontinuation from study treatment.
  Interventions: Drug: Erlotinib; Drug: Second-Line Chemotherapy
- Late Erlotinib (Placebo Comparator): Participants will receive blinded placebo tablets PO once daily in the maintenance setting until disease progression, death, or unacceptable toxicity. Those who demonstrate disease progression may be unblinded to receive second-line erlotinib as 150 mg PO once daily until disease progression, death, or unacceptable toxicity. Participants may be observed during a final SFU period after discontinuation from study treatment.
  Interventions: Drug: Placebo; Drug: Erlotinib

INTERVENTIONS:
Drug: Placebo — Placebo will be administered PO once daily as first-line maintenance until disease progression, death, or unacceptable toxicity.
  Arms: Late Erlotinib
Drug: Erlotinib — Erlotinib will be administered as 150 mg PO once daily until disease progression, death, or unacceptable toxicity, as first-line maintenance or as second-line therapy for those who progress while receiving placebo.
  Other Names: Tarceva
Drug: Second-Line Chemotherapy — Participants who progress on first-line maintenance erlotinib may receive an approved second-line therapy (but not EGFR targeted therapies) until disease progression, death, or unacceptable toxicity. The selected chemotherapy will be non-investigational and chosen at the discretion of the Investigator.
  Arms: Early Erlotinib

SUMMARY:
This double-blind, placebo-controlled study will evaluate the benefit of first-line maintenance erlotinib (Tarceva) versus erlotinib at the time of disease progression in participants with advanced NSCLC who have not progressed following 4 cycles of platinum based-chemotherapy and whose tumor does not harbor an epidermal growth factor receptor (EGFR)-activating mutation. Participants will be randomized to receive either erlotinib 150 milligrams (mg) orally (PO) once daily or placebo. Participants who progress on placebo will receive erlotinib 150 mg PO once daily as second-line therapy, and those who progress on erlotinib may switch to a non-investigational, second-line chemotherapy. Treatments will continue until disease progression, death, or unacceptable toxicity. Participants may also be entered into a final Survival Follow-Up (SFU) period upon treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to (≥) 18 years of age, or legal age of consent if greater than 18
* Advanced or recurrent (Stage IIIB) or metastatic (Stage IV) NSCLC
* Completion of 4 cycles of platinum-based chemotherapy without progression (end of last chemotherapy cycle less than or equal to [≤] 28 days prior to randomization)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Prior exposure to agents directed at human epidermal growth factor receptor (HER) axis (e.g. erlotinib, gefitinib, cetuximab)
* Participants whose tumors harbor an EGFR-activating mutation
* Prior chemotherapy or therapy with systemic anti-neoplastic therapy for advanced disease before Screening
* Use of pemetrexed in maintenance setting (pemetrexed allowed during the chemotherapy run-in)
* Participants who have undergone complete tumor resection after responding to the platinum-based chemotherapy during the Screening phase
* Any other malignancies within 5 years, except for curatively resected carcinoma in situ of the cervix, basal or squamous cell skin cancer, ductal carcinoma in situ, or organ-confined prostate cancer
* Central nervous system (CNS) metastases or spinal cord compression that has not been definitely treated with surgery and/or radiation, or treated CNS metastases or spinal cord compression without stable disease for ≥2 months
* Human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection
* Any inflammatory changes of the surface of the eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (123):
- United States (9):
  - Gilroy, California
  - Washington D.C., District of Columbia
  - Kansas City, Missouri
  - Missoula, Montana
  - Lebanon, New Hampshire
  - Dayton, Ohio
  - Chattanooga, Tennessee
  - Spokane, Washington
  - Tacoma, Washington
- Brazil (6):
  - Belo Horizonte, Minas Gerais
  - Lajeado, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Ijuí, Rondônia
  - Florianópolis, Santa Catarina
  - Santo André, São Paulo
- Bulgaria (6):
  - Gabrovo
  - Haskovo
  - Plovdiv
  - Rousse
  - Sofia
  - Varna
- Canada (4):
  - Windsor, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Regina, Saskatchewan
- China (12):
  - Beijing
  - Changchun
  - Fuzhou
  - Guangzhou
  - Harbin
  - Shanghai
  - Shantou
  - Shenyang
  - Suzhou
  - Tianjin
  - Wuhan
  - Xi'an
- Czechia (6):
  - České Budějovice
  - Jindřichův Hradec
  - Nymburk
  - Ostrava - Poruba
  - Prague
  - Tábor
- France (8):
  - Bayonne
  - Compiègne
  - Gap
  - Libourne
  - Lille
  - Nantes
  - Saint-Brieuc
  - Villefranche-sur-Saône
- Hungary (11):
  - Budapest
  - Deszk
  - Farkasgyepű
  - Győr
  - Gyula
  - Mátraháza
  - Miskolc
  - Székesfehérvár
  - Szolnok
  - Törökbálint
  - Zalaegerszeg
- Italy (10):
  - S. Giovanni Rotondo, Apulia
  - Avellino, Campania
  - Bologna, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Rome, Lazio
  - Legnago, Lombardy
  - Treviglio, Lombardy
  - Livorno, Tuscany
  - Pisa, Tuscany
  - Verona, Veneto
- Latvia (2):
  - Daugavpils
  - Riga
- Lithuania (2):
  - Kaunas
  - Vilnius
- Netherlands (5):
  - Arnhem
  - Heerlen
  - Hoorn
  - Sittard-Geleen
  - Zutphen
- Poland (5):
  - Brzozów
  - Krakow
  - Poznan
  - Wodzisław Śląski
  - Zamość
- Romania (8):
  - Baia Mare
  - Brasov
  - Brăila
  - Bucharest
  - Cluj-Napoca
  - Oradea
  - Ploieşti
  - Târgu Mureş
- Slovakia (6):
  - Banská Bystrica
  - Bardejov
  - Košice
  - Nové Zámky
  - Poprad
  - Rimavská Sobota
- South Africa (4):
  - Cape Town
  - George
  - Port Elizabeth
  - Pretoria
- South Korea (3):
  - Gyeonggi-do
  - Seoul
  - Suwon
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taipei
- Thailand (3):
  - Bangkok
  - Hat Yai
  - Muang
- Ukraine (10):
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kirovograd
  - Kyiv
  - Lutsk
  - Sumy
  - Uzhhorod
  - Vinnytsia
  - Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of three periods: a Blinded Phase (BP), an Open-Label Phase (OLP), and final Survival Follow-Up (SFU). These periods were not necessarily sequential, because the OLP could be "skipped" in select participants. Therefore, the reasons for discontinuation are presented altogether within the Overall Study.
Groups:
- Late Erlotinib: Participants received blinded placebo tablets orally (PO) once daily during the BP in the maintenance setting until disease progression, death, or unacceptable toxicity. Those who demonstrated disease progression were unblinded and could receive second-line erlotinib tablets during the OLP as 150 mg PO once daily, provided by the Sponsor. This treatment continued until disease progression, death, or unacceptable toxicity. If disease progression or unacceptable toxicity occurred during the OLP, the participant entered a final SFU period. Participants could also enter the SFU period directly after the BP if they were unable to receive second-line treatment per protocol.
- Early Erlotinib: Participants received blinded erlotinib tablets, 150 mg PO once daily during the BP in the maintenance setting until disease progression, death, or unacceptable toxicity. Those who demonstrated disease progression were unblinded and could receive an approved second-line therapy (but not epidermal growth factor receptor [EGFR] targeted therapies) or best supportive care (BSC) as chosen by the investigator during the OLP. This treatment continued until disease progression, death, or unacceptable toxicity. If disease progression or unacceptable toxicity occurred during the OLP, the participant entered a final SFU period. Participants could also enter the SFU period directly after the BP if they were unable to receive second-line treatment per protocol.
Period: Overall Study
Arm/Group | Late Erlotinib | Early Erlotinib
Started | 321 | 322
Completed | 0 | 0
Not Completed | 321 | 322
Not completed — Disease Progression | 17 | 14
Not completed — Adverse Event | 2 | 0
Not completed — Death | 243 | 258
Not completed — Lost to Follow-up | 6 | 7
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Study Closed by the Sponsor | 36 | 31
Not completed — Other | 11 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants who were randomized to treatment.
Groups:
- Late Erlotinib: Participants received blinded placebo tablets PO once daily during the BP in the maintenance setting until disease progression, death, or unacceptable toxicity. Those who demonstrated disease progression were unblinded and could receive second-line erlotinib tablets during the OLP as 150 mg PO once daily, provided by the Sponsor. This treatment continued until disease progression, death, or unacceptable toxicity. If disease progression or unacceptable toxicity occurred during the OLP, the participant entered a final SFU period. Participants could also enter the SFU period directly after the BP if they were unable to receive second-line treatment per protocol.
- Early Erlotinib: Participants received blinded erlotinib tablets, 150 mg PO once daily during the BP in the maintenance setting until disease progression, death, or unacceptable toxicity. Those who demonstrated disease progression were unblinded and could receive an approved second-line therapy (but not EGFR targeted therapies) or BSC as chosen by the investigator during the OLP. This treatment continued until disease progression, death, or unacceptable toxicity. If disease progression or unacceptable toxicity occurred during the OLP, the participant entered a final SFU period. Participants could also enter the SFU period directly after the BP if they were unable to receive second-line treatment per protocol.
- Total: Total of all reporting groups
Arm/Group | Late Erlotinib | Early Erlotinib | Total
Number analyzed (Participants) | 321 | 322 | 643
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.1) | 60.8 (8.8) | 60.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 84 | 161
  Male | 244 | 238 | 482

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Died During the Overall Study
Description: Participants were followed for survival until death or premature withdrawal. The percentage of participants who died during the Overall Study (BP, OLP, or SFU) was calculated.
Time Frame: Up to approximately 3.5 years (visits at Baseline and Weeks 6, 12, and 18 and every 12 weeks until/at disease progression during BP; per local standards during OLP; then every 12 weeks during SFU until death)
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Late Erlotinib | Early Erlotinib
Number analyzed (Participants) | 321 | 322
percentage of participants | 73.2 | 75.2

2. Primary Outcome: Overall Survival (OS) as Median Time to Event During the Overall Study
Description: Participants were followed for survival until death or premature withdrawal. OS was defined as the interval between date of randomization and date of death from any cause. Median time to event during the Overall Study (BP, OLP, or SFU) was estimated using the Kaplan-Meier method and expressed in months.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Late Erlotinib | Early Erlotinib
Number analyzed (Participants) | 321 | 322
months | 9.46 [8.38 to 11.33] | 9.72 [8.57 to 11.17]
Statistical Analysis 1: Comparison: Late Erlotinib vs Early Erlotinib; Unstratified Analysis; Test type: Superiority or Other; p = 0.8183, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.85 to 1.22] — The HR and 95% confidence interval (CI) were estimated by Cox regression
Statistical Analysis 2: Comparison: Late Erlotinib vs Early Erlotinib; Stratified Analysis: Stratified according to tumor histology, stage of disease, objective response at Baseline, bevacizumab use, smoking status, and region of enrollment; Test type: Superiority or Other; p = 0.5256, Log Rank; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.87 to 1.32] — The HR and 95% CI were estimated by Cox regression

3. Primary Outcome: Percentage of Participants Event-Free (Alive) at 1 Year During the Overall Study
Description: Participants were followed for survival until death or premature withdrawal. The percentage of participants event-free (i.e., still alive) at 1 year during the Overall Study was calculated.
Time Frame: At 1 year
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Late Erlotinib | Early Erlotinib
Number analyzed (Participants) | 321 | 322
percentage of participants | 41.75 [36.20 to 47.30] | 42.15 [36.60 to 47.70]
Statistical Analysis 1: Comparison: Late Erlotinib vs Early Erlotinib; Test type: Superiority or Other; p = 0.9207, Chi-squared; Difference in Event-Free Rate = -0.40, 95% CI 2-sided [-8.25 to 7.45]

4. Secondary Outcome: Percentage of Participants Who Died or Experienced Disease Progression During Blinded Treatment
Description: Tumor response was evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Disease progression was defined as a greater than or equal to (≥) 20 percent (%) and ≥5-millimeter (mm) increase in the sum of target lesion diameters in reference to the smallest sum on study and/or substantial worsening in non-target disease. The percentage of participants who died or experienced disease progression during the BP was calculated.
Time Frame: Up to approximately 3.5 years (visits at Baseline and Weeks 6, 12, and 18 and every 12 weeks until/at disease progression during BP)
Population: ITT Population.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (Late Erlotinib): Participants received blinded placebo tablets PO once daily during the BP in the maintenance setting until disease progression, death, or unacceptable toxicity.
- Erlotinib (Early Erlotinib): Participants received blinded erlotinib tablets, 150 mg PO once daily during the BP in the maintenance setting until disease progression, death, or unacceptable toxicity.
Arm/Group | Placebo (Late Erlotinib) | Erlotinib (Early Erlotinib)
Number analyzed (Participants) | 321 | 322
percentage of participants | 95.0 | 94.1

5. Secondary Outcome: Progression-Free Survival (PFS) as Median Time to Event During Blinded Treatment
Description: Tumor response was evaluated using RECIST version 1.1. Disease progression was defined as a ≥20% and ≥5-mm increase in the sum of target lesion diameters in reference to the smallest sum on study and/or substantial worsening in non-target disease. PFS was defined as the interval between date of randomization and date of first documented death or disease progression. Median time to event during the BP was estimated using the Kaplan-Meier method and expressed in weeks.
Time Frame: as for outcome 4
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo (Late Erlotinib) | Erlotinib (Early Erlotinib)
Number analyzed (Participants) | 321 | 322
weeks | 12.00 [11.71 to 12.29] | 13.00 [12.14 to 17.43]
Statistical Analysis 1: Comparison: Placebo (Late Erlotinib) vs Erlotinib (Early Erlotinib); Unstratified Analysis; Test type: Superiority or Other; p = 0.4759, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.80 to 1.11] — The HR and 95% CI were estimated by Cox regression
Statistical Analysis 2: Comparison: Placebo (Late Erlotinib) vs Erlotinib (Early Erlotinib); [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1635, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.72 to 1.06] — The HR and 95% CI were estimated by Cox regression

6. Secondary Outcome: Percentage of Participants Event-Free (Alive and No Disease Progression) at 6 Months During Blinded Treatment
Description: Tumor response was evaluated using RECIST version 1.1. Disease progression was defined as a ≥20% and ≥5-mm increase in the sum of target lesion diameters in reference to the smallest sum on study and/or substantial worsening in non-target disease. The percentage of participants event-free (i.e., still alive and without disease progression) at 6 months during the BP was calculated.
Time Frame: At 6 months
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Late Erlotinib) | Erlotinib (Early Erlotinib)
Number analyzed (Participants) | 321 | 322
percentage of participants | 24.22 [19.50 to 28.94] | 27.11 [22.19 to 32.02]
Statistical Analysis 1: Comparison: Placebo (Late Erlotinib) vs Erlotinib (Early Erlotinib); Test type: Superiority or Other; p = 0.4069, Chi-squared; Difference in Event-Free Rate = -2.89, 95% CI 2-sided [-9.70 to 3.93]

7. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) According to RECIST During Blinded Treatment
Description: Tumor response was evaluated using RECIST version 1.1. CR was defined as disappearance of all target and non-target lesions and short-axis reduction to less than (<) 10 mm of any pathological lymph nodes. PR was defined as a ≥30% decrease in the sum of target lesion diameters in reference to the Baseline sum. The percentage of participants with a best overall response of either CR or PR (i.e., the objective response rate [ORR]) during the BP was calculated, and corresponding 95% CI was constructed using the Pearson-Clopper method.
Time Frame: as for outcome 4
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Late Erlotinib) | Erlotinib (Early Erlotinib)
Number analyzed (Participants) | 321 | 322
percentage of participants | 3.7 [1.95 to 6.44] | 6.5 [4.08 to 9.80]
Statistical Analysis 1: Comparison: Placebo (Late Erlotinib) vs Erlotinib (Early Erlotinib); Test type: Superiority or Other; p = 0.1097, Chi-squared; Difference in Response Rate = 2.78, 95% CI 2-sided [-0.78 to 6.35] — The 95% CI for difference in response rates was constructed using the Anderson-Hauck method
Statistical Analysis 2: Comparison: Placebo (Late Erlotinib) vs Erlotinib (Early Erlotinib); Test type: Superiority or Other; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.87 to 3.72] — The 95% CI for OR was constructed using the Wald method

8. Secondary Outcome: Percentage of Participants by Best Overall Response According to RECIST During Blinded Treatment
Description: Tumor response was evaluated using RECIST version 1.1. CR was defined as disappearance of all target and non-target lesions and short-axis reduction to <10 mm of any pathological lymph nodes. PR was defined as a ≥30% decrease in the sum of target lesion diameters in reference to the Baseline sum. Stable disease (SD) was defined as neither sufficient shrinkage in target lesions to qualify for PR nor sufficient growth to qualify for disease progression. Disease progression (progressive disease/PD) was defined as a ≥20% and ≥5-mm increase in the sum of target lesion diameters in reference to the smallest sum on study and/or substantial worsening in non-target disease. The percentage of participants with each level of best tumor response during the BP was calculated, and corresponding 95% CI was constructed using the Pearson-Clopper method.
Time Frame: as for outcome 4
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Late Erlotinib) | Erlotinib (Early Erlotinib)
Number analyzed (Participants) | 321 | 322
percentage of participants
  CR | 0.6 [0.08 to 2.23] | 0.9 [0.19 to 2.70]
  PR | 3.1 [1.50 to 5.65] | 5.6 [3.35 to 8.69]
  SD | 55.5 [49.83 to 60.97] | 54.7 [49.04 to 60.19]
  PD | 38.6 [33.27 to 44.20] | 32.3 [27.22 to 37.71]
  Missing | 2.2 [0.88 to 4.44] | 6.5 [4.08 to 9.80]

9. Secondary Outcome: Percentage of Participants With CR, PR, or SD According to RECIST During Blinded Treatment
Description: Tumor response was evaluated using RECIST version 1.1. CR was defined as disappearance of all target and non-target lesions and short-axis reduction to <10 mm of any pathological lymph nodes. PR was defined as a ≥30% decrease in the sum of target lesion diameters in reference to the Baseline sum. SD was defined as neither sufficient shrinkage in target lesions to qualify for PR nor sufficient growth to qualify for disease progression. The percentage of participants with a best overall response of CR, PR, or SD (i.e., the disease control rate [DCR]) during the BP was calculated, and corresponding 95% CI was constructed using the Pearson-Clopper method.
Time Frame: as for outcome 4
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Late Erlotinib) | Erlotinib (Early Erlotinib)
Number analyzed (Participants) | 321 | 322
percentage of participants | 59.2 [53.59 to 64.62] | 61.2 [55.62 to 66.53]
Statistical Analysis 1: Comparison: Placebo (Late Erlotinib) vs Erlotinib (Early Erlotinib); Test type: Superiority or Other; p = 0.6062, Chi-squared; Difference in Response Rate = 1.99, 95% CI 2-sided [-5.74 to 9.72] — The 95% CI for difference in response rates was constructed using the Anderson-Hauck method
Statistical Analysis 2: Comparison: Placebo (Late Erlotinib) vs Erlotinib (Early Erlotinib); Test type: Superiority or Other; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.79 to 1.49] — The 95% CI for OR was constructed using the Wald method

ADVERSE EVENTS:
Time Frame: Up to approximately 4.5 years (visits at Baseline and Weeks 6, 12, and 18 and every 12 weeks until disease progression, death, or unacceptable toxicity during BP; per local standards and 28 days after last visit during OLP)
Description: Safety Population: All participants who received at least one dose of study treatment, according to drug actually received. Non-serious adverse events (NSAEs) were not collected in the OLP. Hence, 0 participants would be affected and at risk in "Other (Not Including Serious) Adverse Events". However, an NSAE in 1 participant was reported to Roche outside protocol (see "Rash"). Other NSAEs that may have occurred during the OLP are not included in the table because they were not reported to Roche.
Groups:
- Second-Line Erlotinib (Late Erlotinib): Participants who received blinded placebo and who demonstrated disease progression were unblinded and could receive second-line erlotinib as 150-mg tablets PO once daily, provided by the Sponsor. This treatment continued during the OLP until disease progression, death, or unacceptable toxicity.
- Second-Line Chemotherapy (Early Erlotinib): Participants who received blinded erlotinib and who demonstrated disease progression were unblinded and could receive an approved second-line therapy (but not EGFR targeted therapies) or BSC as chosen by the investigator. This treatment continued during the OLP until disease progression, death, or unacceptable toxicity.
Arm/Group | Placebo (Late Erlotinib) | Erlotinib (Early Erlotinib) | Second-Line Erlotinib (Late Erlotinib) | Second-Line Chemotherapy (Early Erlotinib)
Serious Adverse Events (participants affected / at risk) | 27/319 | 36/322 | 23/248 | 8/162
Other Adverse Events (participants affected / at risk) | 107/319 | 206/322 | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Late Erlotinib) (N=319) | Erlotinib (Early Erlotinib) (N=322) | Second-Line Erlotinib (Late Erlotinib) (N=248) | Second-Line Chemotherapy (Early Erlotinib) (N=162)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Pneumonia (Infections and infestations) | 3 | 4 | 2 | 1
Abscess oral (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorroids thrombosed (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 1 | 0
Perforated ulcer (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Finger amputation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Meningeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (Late Erlotinib) (N=319) | Erlotinib (Early Erlotinib) (N=322) | Second-Line Erlotinib (Late Erlotinib) (N=1) | Second-Line Chemotherapy (Early Erlotinib) (N=0)
Diarrhoea (Gastrointestinal disorders) | 14 | 78 | 0/0 | 0
Chest pain (General disorders) | 11 | 17 | 0/0 | 0
Fatigue (General disorders) | 20 | 21 | 0/0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 11 | 21 | 0/0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 31 | 0/0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 27 | 0/0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 17 | 0/0 | 0
Rash (Skin and subcutaneous tissue disorders) | 32 | 127 | 1 | 0 — Per protocol, NSAEs were not collected in the OLP. However, an NSAE in 1 participant in the "Second-Line Erlotinib (Late Erlotinib)" arm was reported outside protocol and coded with MedDRA (18.1). As such, this single event is presented in the table.
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 17 | 0/0 | 0

LIMITATIONS AND CAVEATS:
Following the final analysis, the study was closed and all remaining participants were withdrawn from the study and considered "Not Completed" (as presented in the Participant Flow). However, the overall status of study was confirmed as completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.